CLINICAL TRIAL: NCT01276847
Title: A Clinical Trial to Assess the Effects of Ustekinumab and Etanercept on Skin and Blood Biomarkers of Psoriasis in Patients With Moderate to Severe Disease
Brief Title: A Study to Assess the Effect of Ustekinumab (Stelara®) and Etanercept (Enbrel®) in Participants With Moderate to Severe Psoriasis (MK-0000-206)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0000-206
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Results first posted 2013-02-28 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Psoriasis
Keywords: psoriasis; Ustekinumab; Stelara; Etanercept; Enbrel
MeSH Terms: conditions — Psoriasis | interventions — Ustekinumab; Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ustekinumab (Experimental)
  Interventions: Drug: Ustekinumab
- Etanercept (Active Comparator)
  Interventions: Drug: Etanercept
- No treatment (No Intervention)

INTERVENTIONS:
Drug: Ustekinumab — Ustekinumab 45 mg per dose, administered subcutaneously for participants weighing ≤ 100 kg, and ustekinumab 90 mg per dose administered subcutaneously for participants weighing > 100 kg on Day 1, and Weeks 4 and 16
  Other Names: Stelara
  Arms: Ustekinumab
Drug: Etanercept — Etanercept 50 mg twice weekly by self-administered subcutaneous injection for 12 weeks, then once weekly for 4 weeks
  Other Names: Enbrel
  Arms: Etanercept

SUMMARY:
This is a two-part study. The purpose of the pilot study (Part 1) is to optimize the acquisition, handling and shipping procedure for skin biopsies obtained from participants with plaque psoriasis. No treatment will be administered. Part 2 will include 2 cohorts. In Cohort 1, the effects of 16 weeks of treatment with either ustekinumab or etanercept on biomarkers in lesional skin in participants with moderate to severe psoriasis will be evaluated. In Cohort 2, biomarkers of lesional skin from participants with moderate to severe psoriasis who are not treated with biologic therapy will be evaluated over 16 weeks. The primary hypothesis is that treatment with ustekinumab reduces messenger RNA (mRNA) expression of genes in the interleukin 12 (IL-12) pathway that are modulated by interferon gamma (IFN-γ).

ELIGIBILITY:
Inclusion Criteria:

* Is unlikely to conceive (for female participants of reproductive potential)- Part 2
* Has a diagnosis of predominantly plaque psoriasis for ≥ 6 months-Parts 1 and 2
* Has a plaque-type psoriatic lesion with a Target Lesion Score (TLS) score of ≥ 6 in a hidden area of the body such as the abdomen, thighs, lower back or buttock that is suitable for biopsy- Part 1
* Is considered to be a candidate for phototherapy or systemic therapy - Part 2
* Has a Psoriasis Area and Severity Index (PASI) score ≥ 12 at Baseline - Part 2
* Has psoriasis body surface area (BSA) involvement ≥ 10% at Baseline - Part 2
* Has a Physician's Global Assessment (PGA) of at least moderate disease (moderate, marked, or severe) at Baseline - Part 2
* Is considered to be eligible according to the tuberculosis (TB) screening criteria - Part 2

Exclusion Criteria:

* Has nonplaque forms of psoriasis specifically erythrodermic psoriasis, predominantly pustular psoriasis, medication-induced or medication-exacerbated psoriasis, or new onset guttate psoriasis - Parts 1 and 2
* Women of childbearing potential who are pregnant, intend to become pregnant (within 6 months of completing the trial), or are lactating - Parts 1 and 2
* Has a history of neoplastic disease or concurrent malignancy - Part 2
* Requires oral or injectable corticosteroids during the trial - Part 2
* Have any infection requiring treatment with antibiotics within 2 weeks prior to screening or serious infection requiring hospitalization or treatment with IV antibiotics within 8 weeks prior to screening - Part 2
* Has a positive human immunodeficiency virus (HIV) test result, hepatitis B surface antigen, or hepatitis C test result - Part 2
* Has received live virus vaccination within 4 weeks prior to screening or who intends to receive live virus vaccination during the trial - Part 2
* Has previous exposure to any agents targeting IL-12 and/or IL-23 (e.g. ustekinumab) - Part 2
* Has prior exposure tumor necrosis factor (TNF) antagonists (e.g. infliximab, etanercept, golimumab, adalimumab) and discontinued due to lack of efficacy or for adverse effects - Part 2
* Has been treated with any medications that are associated with Progressive Multifocal Leukoencephalopathy (PML), such as efalizumab (Raptiva) or natalizumab (Tysabri) - Part 2
* Has taken any immunosuppressive agents (e.g. corticosteroids, methotrexate, azathioprine, cyclosporine) for treatment of conditions other than for Psoriasis within 4 weeks of screening - Part 2
* Is currently taking any of the prohibited medications and is unwilling to washout of the medication(s) for the indicated timeframe prior to screening and for the duration of the study - Part 2

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept: Etanercept : Etanercept 50 mg twice weekly by self-administered subcutaneous injection for 12 weeks, then once weekly for 4 weeks
- No Treatment: No treatment administered
- Ustekinumab: Ustekinumab : Ustekinumab 45 mg per dose, administered subcutaneously for participants weighing ≤ 100 kg, and ustekinumab 90 mg per dose administered subcutaneously for participants weighing > 100 kg on Day 1, and Weeks 4 and 16
Period: Overall Study
Arm/Group | Etanercept | No Treatment | Ustekinumab
Started | 10 | 10 | 20
Completed | 9 | 10 | 20
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etanercept | No Treatment | Ustekinumab | Total
Number analyzed (Participants) | 10 | 10 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (12.5) | 53.4 (13.0) | 45.7 (12.1) | 46.1 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 7 | 12
  Male | 6 | 9 | 13 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Composite Gene Expression Score Based on IL-12 Pathway Related Interferon Gamma (IFN-γ)-Modulated Genes in Psoriatic Lesions of Participants Treated With Ustekinumab
Description: Skin biopsies were collected from participants at baseline and after treatment with ustekinumab for 1,2,4 and 16 weeks. The expression of messenger RNA (mRNA) from three pre-defined IL-12 pathway related genes, modulated by interferon gamma (IFN-γ), namely IFN-γ, inducible nitric oxide synthase(iNOS) and CXC motif chemokine 10(CXCL10) was quantitated by real-time polymerase chain reaction (qPCR), with the data normalized by the delta-delta Ct method. The expression score for each gene, showing the percentage difference from baseline, was calculated as follows : [(baseline - post baseline)/baseline] x 100. Composite gene expression scores were derived for each individual by summing the expression scores of the individual genes. Positive composite scores denote a decrease from baseline in gene expression.
Time Frame: Baseline and Weeks 1, 2, 4, and 16
Population: Pre-specified to be collected only in participants treated with Ustekinumab. One participant treated with Ustekinumab with extreme outlying data, likely due to mislabeling of lesional and nonlesional tissues, was excluded from the analysis.
Measure: Median (90% Confidence Interval); unit: Gene expression score
Arm/Group | Ustekinumab
Number analyzed (Participants) | 19
Gene expression score
  Week 1 | 53.68 [19.90 to 96.34]
  Week 2 | 130.54 [38.47 to 158.00]
  Week 4 | 180.19 [130.50 to 189.38]
  Week 16 | 240.29 [139.44 to 257.76]
Statistical Analysis 1: Comparison: Ustekinumab; Week 1; Test type: Superiority or Other; p = 0.016, Wilcoxon (Mann-Whitney) — unadjusted 1-sided p-value, α = 0.05; One-sample test
Statistical Analysis 2: Comparison: Ustekinumab; Week 2; Test type: Superiority or Other; p = 0.007, Wilcoxon (Mann-Whitney) — unadjusted 1-sided p-value, α = 0.05; One-sample test
Statistical Analysis 3: Comparison: Ustekinumab; Week 4; Test type: Superiority or Other; p = 0.00015, Wilcoxon (Mann-Whitney) — unadjusted 1-sided p-value, α = 0.05; One-sample test
Statistical Analysis 4: Comparison: Ustekinumab; Week 16; Test type: Superiority or Other; p = 0.000184, Wilcoxon (Mann-Whitney) — unadjusted 1-sided p-value, α = 0.05; One-sample test

2. Secondary Outcome: Change From Baseline in Composite Gene Expression Score Based on Interleukin 23 (IL-23) Pathway Related Genes in Psoriatic Lesions of Participants Treated With Ustekinumab
Description: Skin biopsies were collected from participants at baseline and after treatment with ustekinumab for 1,2,4 and 16 weeks. The mRNA expression of eight pre-defined IL-23 pathway related genes, namely beta 4 defensin (DEFB4), CXC motif chemokine 8 (CXCL8), Interleukins 17A, 17F, 20, 22, 23A (IL-17, IL-17F, IL-20, IL-22, IL-23A) and cyclic AMP dependent protein kinase (CAMP) was quantitated by qPCR, with the data normalized by the delta-delta Ct method. The expression score for each gene, showing the percentage difference from baseline, was calculated as follows : [(baseline - post baseline)/baseline] x 100. Composite gene expression scores were derived for each individual by summing the expression scores of the individual genes. Positive composite scores denote a reduction from baseline in gene expression.
Time Frame: Baseline and Weeks 1, 2, 4, and 16
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: Gene expression score
Arm/Group | Ustekinumab
Number analyzed (Participants) | 19
Gene expression score
  Week 1 | 44.24 [-170.81 to 185.43]
  Week 2 | 399.31 [96.66 to 442.98]
  Week 4 | 412.79 [304.55 to 550.96]
  Week 16 | 716.14 [358.51 to 746.78]
Statistical Analysis 1: Comparison: Ustekinumab; Week 1; Test type: Superiority or Other; p = 0.397, Wilcoxon (Mann-Whitney) — unadjusted 1-sided p-value, α = 0.05; One-sample test
Statistical Analysis 2: Comparison: Ustekinumab; Week 2; Test type: Superiority or Other; p = 0.010, Wilcoxon (Mann-Whitney) — unadjusted 1-sided p-value, α = 0.05; One-sample test
Statistical Analysis 3: Comparison: Ustekinumab; Week 4; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney) — unadjusted 1-sided p-value, α = 0.05; One-sample test
Statistical Analysis 4: Comparison: Ustekinumab; Week 16; Test type: Superiority or Other; p = 0.000215, Wilcoxon (Mann-Whitney) — unadjusted 1-sided p-value, α = 0.05; One-sample test

3. Secondary Outcome: Change From Baseline in Gene Expression Score for Interleukin 17 (IL-17) in Psoriatic Lesions of Participants Treated With Etanercept
Description: Participants had skin biopsies performed at baseline and after treatment with etanercept for 1,2,4 and 16 weeks. The expression of IL-17 mRNA was quantitated by qPCR, with the data normalized by the delta-delta Ct method. The expression score, showing the percentage difference from baseline, was calculated as follows : [(baseline - post baseline)/baseline] x 100.
Time Frame: Baseline and Weeks 1, 2, 4, and 16
Population: Pre-specified to be collected only in participants treated with Etanercept.
Measure: Median (90% Confidence Interval); unit: Gene expression score
Arm/Group | Etanercept
Number analyzed (Participants) | 10
Gene expression score
  Week 1 | 5.17 [-118.88 to 15.68]
  Week 2 | 17.75 [-154.28 to 44.76]
  Week 4 | 65.50 [-10.94 to 84.78]
  Week 16 | 52.77 [-24.74 to 91.70]
Statistical Analysis 1: Comparison: Etanercept; Week 1; Test type: Superiority or Other; p = 0.787, Wilcoxon (Mann-Whitney) — unadjusted 1-sided p-value, α = 0.05; One-sample test
Statistical Analysis 2: Comparison: Etanercept; Week 2; Test type: Superiority or Other; p = 0.577, Wilcoxon (Mann-Whitney) — unadjusted 1-sided p-value, α = 0.05; One-sample test
Statistical Analysis 3: Comparison: Etanercept; Week 4; Test type: Superiority or Other; p = 0.053, Wilcoxon (Mann-Whitney) — unadjusted 1-sided p-value, α = 0.05; One-sample test
Statistical Analysis 4: Comparison: Etanercept; Week 16; Test type: Superiority or Other; p = 0.098, Wilcoxon (Mann-Whitney) — unadjusted 1-sided p-value, α = 0.05; One-sample test

ADVERSE EVENTS:
Arm/Group | Etanercept | No Treatment | Ustekinumab
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10 | 0/20
Other Adverse Events (participants affected / at risk) | 3/10 | 2/10 | 6/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=10) | No Treatment (N=10) | Ustekinumab (N=20)
Foetal Distress Syndrome (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=10) | No Treatment (N=10) | Ustekinumab (N=20)
Vitreous Detachment (Eye disorders) | 0 | 1 | 0
Cyst (General disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 3
Pharyngitis Streptococcal (Infections and infestations) | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 2
Procedural Site Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Gestational Diabetes (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.